CLINICAL TRIAL: NCT04857294
Title: Unilateral TMJ Discectomy Without Interposal Material in Patients With Disc Perforation or Fragmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Portugues da Face (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMJDISCECT
Record Dates: First submitted 2021-04-10; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Temporomandibular Disorders
Keywords: Temporomandibular; TMJ Discectomy; TMJ Meniscectomy; TMJ Surgery
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discectomy (Experimental): Unilateral Discectomy
  Interventions: Procedure: TMJ unilateral discectomy

INTERVENTIONS:
Procedure: TMJ unilateral discectomy — All patients underwent general anesthesia with nasotracheal intubation, managed in most cases with intravenous anesthesia protocol, usually with remifentanil infusion. Intraoperative steroids, usually dexamethasone, were administered primarily to minimize postoperative swelling. A classic preauricular incision or a root of helix inter tragus notch incision (RHITNI) was used in most cases, as previously described. No bandage or special care was performed after the surgery. No air washing restrictions were recommended.

SUMMARY:
Temporomandibular joint (TMJ) discectomy is one of the most popular surgical techniques for painful TMJ. Previous studies have demonstrated predictable results of discectomy with optimal results in pain reduction and maximum mouth opening (MMO) improvement. However, those studies had most of the times varied inclusion criteria. A 4-year prospective study was designed including patients treated with unilateral TMJ discectomy without interposal material as the first surgical procedure for two specific intra-articular diagnosis: disc perforation and disc fragmentation.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are the most prevalent orofacial pain source of nondental origin. Those disorders can be due to a heterogeneous group of pathologies affecting the temporomandibular joint (TMJ), the jaw muscles, or both. TMD symptoms prevalence has been reported between 10 to 33% of the population. The most common symptoms include pain, joint sounds, limitation of mandibular movement, facial deformities, condyle dislocation and recurrent headaches. These symptoms can negatively affect the quality of life. Surgical treatments for TMD are reserved for specific cases, however with the popularization of mini-invasive surgical techniques such as TMJ arthroscopy, more patients have been eligible for these mini-invasive techniques, amplifying the scope of TMJ surgery. In diagnostics such as ankylosis, tumors and growth abnormalities, TMJ open surgery is strongly recommended. However, those diagnosis and relatively uncommon. TMJ internal derangement involving disc position/integrity and osteoarthrosis are more frequent, but the surgical indication is relative.

From all the open surgery techniques, TMJ discectomy without interposal material is probably one of the most popular procedures. Recently, was showed that bilateral discectomy can induce severe TMJ changes detected with both imaging and histopathologic analysis in black Merino sheep. Besides, the critical histological and imaging results, functional masticatory alterations were not influenced by TMJ degenerative changes. Also, in other preclinical study, disc and fibrocartilage removal lead to traumatic TMJ ankylosis. It is interesting to observe the role of the condyle and temporal fibrocartilage, balancing the disc function. In humans, short-term studies on TMJ discectomy were associated with good results. In fact, in other retrospective study was showed discectomy without replacement is effective improving the preoperative maximum mouth opening (MMO). Despite the good clinical outcome, some studies have observed degenerative changes in imaging analysis. Together, clinical and preclinical results showed TMJ discectomy is a suboptimal technique, and an effective disc substitute, acting as a cushion between the condyle and temporal fossa could, in theory, improve these results. Despite extensive research in the field of tissue engineering, currently no appropriate disc substitute has demonstrated safety and efficacy. In fact, the last guidelines do not recommend disc replacement because nonvalid option showed superiority over discectomy alone. While there is no effective disc substitute, discectomy is often used when the disc is partial or total damaged and cannot be salvaged and/or and when symptoms fail to improve with other techniques. The inclusion criteria heterogeneity in previous studies, retrospective studies and non-randomization makes it difficult to draw clear conclusions about this technique. The investigators designed a rigorous prospective study for patients with: 1) unilateral TMJ disc perforation or 2) unilateral TMJ disc fragmentation. Those patients were proposed to unilateral TMJ discectomy. Most of the times, when the disc is damaged, the bone fibrocartilage is distorted and the authors wanted to understand the role of discectomy is those patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old;
* Unilateral TMJ pain >7 (0-10 VAS) and/or MMO < 30mm;
* MRI presenting unilateral disc perforation or disc fragmentation
* Clinical and imaging examination with criteria for unilateral TMJ discectomy

Exclusion Criteria:

* Previous TMJ surgical intervention;
* Concomitant contralateral surgery;
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analogue Scale (0,10) | Pre-surgery
  VAS, 0-10, with 0 being no pain and 10 having maximum unbearable pain
Pain (Visual Analogue Scale (0,10) | Through study completion, an average of 2 years
  VAS, 0-10, with 0 being no pain and 10 having maximum unbearable pain

SECONDARY OUTCOMES:
Maximum mouth opening (MMO, mm) | Pre-surgery
  Mouth opening measured with a ruler (mm)
Maximum mouth opening (MMO, mm) | Through study completion, an average of 2 years
  Mouth opening measured with a ruler (mm)
Muscle tenderness (0-3 scale) | Pre-surgery
  0-3, corresponding to a muscle tenderness scale in masseter and temporalis muscle (0-whithout muscle tenderness, 3 - maximum muscle tenderness)
Muscle tenderness (0-3 scale) | Through study completion, an average of 2 years
  0-3, corresponding to a muscle tenderness scale in masseter and temporalis muscle (0-whithout muscle tenderness, 3 - maximum muscle tenderness)

CONTACTS AND LOCATIONS:
Overall Officials: David Ângelo, MD, PhD, Study Director — Instituto Português da Face
Locations (1):
- Instituto Português da Face, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No